CLINICAL TRIAL: NCT06780358
Title: Study of bladdeR Cancer Detection in Standard White Light Versus AI-Supported Endoscopy-02
Acronym: RAISE02
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cystotech (Industry)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RAISE02-24-02
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Premarket Confirmatory, National, single-center, randomized, prospective, non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WLC detection (No Intervention): Detection of bladder cancer is conducted according to state-of-the-art procedures in white light modality.
- AI model - WLC supported detection (Experimental): Detection of bladder cancer in white light supported by a pre-market AI-support tool.
  Interventions: Device: AI supported detection of bladder cancer

INTERVENTIONS:
Device: AI supported detection of bladder cancer — AI-model-supported detection of bladder cancer during white light cystoscopy
  Arms: AI model - WLC supported detection

SUMMARY:
This study is being conducted to investigate if an artificial intelligence support tool is non-inferior in detecting bladder cancer compared to the traditional method, standard white light cystoscopy (WLC). The researchers will compare how well the artificial intelligence tool and WLC perform in detecting bladder cancer through a controlled, organized testing process.

DETAILED DESCRIPTION:
This clinical investigation aims to confirm that an artificial intelligence model utilizing a Convolutional Neural Network (CNN) can achieve sensitivity in detecting bladder cancer that is non-inferior to traditional white light cystoscopy (WLC) in a randomized controlled trial. The investigational artificial intelligence device leverages the advanced capabilities of CNNs, a type of deep learning model designed to analyze visual imagery with high precision.

ELIGIBILITY:
Inclusion Criteria:

* Men and women adults, age >18 years old

Suspicion of primary or recurrent bladder cancer

Willingness to sign the Informed Consent Form (ICF) for the CI

Ability to comprehend the oral and written Patient Information Leaflet (PIL)

Exclusion Criteria:

* Not able or willing to sign the Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of standard WLC compared to WLC assisted by the AI model evaluated with a non-inferiority margin of 5%. | 7 month
  To determine whether the AI model is non-inferior with regards to sensitivity compared to standard WLC in a randomized controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jakobsen, Principal Investigator — Department of Urology, Aarhus University Hospital, denmark
Locations (1):
- Department of Urology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Sharing the IPD conflicts with the collaboration agreement.